CLINICAL TRIAL: NCT06286111
Title: Red Cell Distribution Width as a Predictor for Post Operative Atrial Fibrillation After Open Heart Surgeries
Brief Title: Red Cell Distribution Width as a Predictor for Post Operative Atrial Fibrillation After Open Heart Surgries
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: ASU MD
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Inflammatory Marker; Heart; Surgery, Heart, Functional Disturbance as Result
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

SUMMARY:
In this study we investigate the correlation between RDW and POAF, as we use the RDW as a predictor for inflammation for prediction of POAF

DETAILED DESCRIPTION:
In this study we investigate the relation between Red Cell Distribution Width and post operative atrial fibrillation after open heart surgery as it's a major complication with high incidence, this complication prolong the in hosoital stay, postulated mechanism of Post Operative Atrial Fibrillation that it's due to inflammation and oxidative stress, after applying specific inclusion and exclusion criteria, recording the preoperative labs including RDW and follow up patients 48 hours post operative in the ICU and recording post operative labs and ECG, and compare the RDW of patients developed POAF and patients who didn't develop POAF

ELIGIBILITY:
Inclusion Criteria:

* Female or Male patient with range of age 35-65 years
* Elective Cardiac surgery
* Cardiopuomonary bypass machine used
* Normal Sinus Rhythm

Exclusion Criteria:

* Echo showing left atrial diameter above 4 cm
* Patient on rythm control medications
* Patient undergoing emergency surgery
* History of cardiac Tachyarrhythemia

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing open heart surgery with cardiopulmonary bypass used intraoperative, with no history of cardiac tachyarrythemia and not using rythm control drugs with normal cardiac dimensions
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Red cell distribution width as a predictor for Post-operative Atrial fibrillation after Open Heart Surgeries | 48 hours post operative
  The correlation between Red cell distribution width and post operative atrial fibrillation after open heart sutgeries

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams University, Cairo, Egypt